CLINICAL TRIAL: NCT07172243
Title: BE.Amycon Biobank & Data Registry UZ Leuven: Human Body Material (HBM) Collection and Data Collection of Patients With Amyloidosis
Brief Title: BE.Amycon Biobank & Data Registry UZ Leuven
Status: Not yet recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: BE.AMYCON_UZL_WP2_02
Record Dates: First submitted 2025-08-20; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Amyloidosis; AL Amyloidosis; Amyloidosis Cardiac
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, biopsy (in the context of amyloidosis), subcuteanous fat aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to collect and store human body material (HBM) of patients with amyloidosis in a biobank "BE.Amycon biobank" for future research and to collect clinical data of patients with amyloidosis in a database "BE.Amycon data registry".

DETAILED DESCRIPTION:
With the support of VIB (Vlaams Instituut voor Biotechnologie) Grand Challenges Program, this project aims to establish the BElgian AMYloidosis CONsortium (BE.AMYCON) by joining forces of VIB researchers, a state-of-the-art diagnostic platform, and clinicians from various disciplines and different institutes. Such a consortium will address patient needs and improve outcomes on many levels.

The aim is is to establish a GDPR (General Data Protection Regulation)-proof HBM biobank in the context of amyloidosis. HBM of patients with suspected or confirmed amyloidosis will be prospectively collected and stored for future scientific research. In addition to the HBM collection, a database with personal and health data of patients diagnosed with amyloidosis (any subtype) will be established in order to get better insights on the disease presentation, disease evolution pattern, treatment plans and responses and survival.

ELIGIBILITY:
Inclusion Criteria:

* Provide consent and sign informed consent form
* Age 18 years or older
* Diagnosis of amyloidosis (suspected or confirmed, any subtypes)
* For the prospective sample collection only: newly diagnosed (any subtype) or at relapse (AL amyloidosis)

Exclusion Criteria:

* Not willing to sign informed consent
* Not able to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with amyloidosis
Sampling Method: Probability Sample
Enrollment: 505 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of a data registry: participant baseline demographics | Baseline
  Demographic characteristics of amyloidosis participants will be assessed at baseline.
Establishment of a data registry: description of the disease characteristics of patients with amyloidosis at diagnosis | Baseline
  Disease characteristics of amyloidosis (disease presentation and symptoms, type of organ involvment, results of diagnostic tests (lab values, imaging, biopsy)) will be collected at moment of diagnosis.
Establishment of a data registry: treatment in participants with amyloidosis | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  Description of treatment (type of treatment per line of treatment) of participants with amyloidosis within routine clinical care.
Establishment of a biobank with biological samples (blood, urine, tissue) from patients with amyloidosis | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 2 years
  Biological samples (blood, urine, tissue) will be collected from patients with amyloidosis.

SECONDARY OUTCOMES:
Best Response | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  Documentation of response rates per line of treatment
Duration of response | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years.
  Duration of response is defined as the time from the date of initial documentation of a response to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death.
Time to Next Treatment (TTNT) | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years.
  TTNT is defined as the time from the date of initiation of regimen to the initiation of next regimen for each successive therapy received.
Overall Survival (OS) | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  OS is defined as the time from the date of initiation of therapy to the date of death from any cause (or last documented follow-up).
Progression-free survival (PFS) | From enrollment of the patient until death, until loss to follow-up or withdrawal of informed consent, whichever comes first, up to 10 years
  PFS is defined as the time from the date of initiation of therapy to the date of progression or death of any cause, whichever occurs first (or last documented follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delforge, Principal Investigator — UZ Leuven Gasthuisberg
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon signed MTA and DTA and approval by steering committee meeting and ethics committee.
Time Frame: Per approved user protocol
Access Criteria: upon signed MTA and DTA and approval by steering committee meeting and ethics committee